CLINICAL TRIAL: NCT01209650
Title: Expanded Access Program BIBW 2992 for Non Small Cell Lung Cancer ( NSCLC) Last Line Treatment
Brief Title: LUX Lung Special Access Scheme Australia Named Patient Use (NPU)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.47
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

INTERVENTIONS:
Drug: BIBW 2992 — tablets

SUMMARY:
The program will provide early access to the investigational drug BIBW 2992 to treat patients with advanced NSCLC who have failed at least 12 weeks on erlotinib or gefitinib.

The Compassionate Use Programme will also provide additional safety and efficacy information on BIBW 2992 use.

Named Patient Use (NPU)

ELIGIBILITY:
Inclusion criteria:

* Patients with pathologic confirmation of adenocarcinoma of the lung Stage IIIB with pleural effusion or Stage IV

Exclusion criteria:

* Brain metastases which are symptomatic; patients with treated, asymptomatic brain metastases are eligible with stable brain disease for at least four 4 weeks without the requirement for steroids or anti epileptic therapy
* Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom as judged by the investigator.
* Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator, would either compromise patient safety or interfere with the evaluation of the safety of the test drug
* History of cardiac disease that is clinically significant, as judged by the investigator or uncontrolled cardiac disease (including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association (NYHA) functional classification of 3)
* Cardiac left ventricular function with resting ejection fraction of less than 50%
* Bilirubin 1.5 mg / dl (26 mol / L, SI unit equivalent)
* Aspartate amino transferase (AST) or alanine amino transferase (ALT) three times the upper limit of normal (if related to liver metastases five times the upper limit of normal)
* Serum creatinine 1.5 times of the upper normal limit or calculated/measured creatine clearance 45ml/min
* Women of child-bearing potential or men who are able to father a child unwilling to use a medically acceptable method of contraception during the trial
* Pregnancy or breast feeding
* Patients unable to comply with the protocol
* Patients with known HIV, active hepatitis B or active hepatitis C
* Pre-existing Interstitial Lung Disease (ILD)
* Requirement for treatment with any of the prohibited concomitant medications listed in Section 4.2.2.1.
* Patients already pre-treated with BIBW 2992

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1200.47.1 Boehringer Ingelheim Investigational Site, North Ryde, New South Wales, Australia